CLINICAL TRIAL: NCT03610789
Title: A Multicenter, Post-Market Clinical Follow-up Study of Subjects With the REDAPT™ System Monolithic Sleeveless/Sleeved Stem and/or Fully Porous Acetabular Shell With XLPE Liner and/or Modular Shell Components Previously Implanted
Status: Enrolling by invitation | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REDAPT 17-4538-02
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- REDAPT Revision Femoral System: REDAPT Revision Femoral System Monolithic Sleeveless Stems, monolithic sleeved stems and/or Acetabular Components or modular shells and/or augments
  Interventions: Device: REDAPT

INTERVENTIONS:
Device: REDAPT — REDAPT Monolithic Sleeveless Stems and Acetabular Cup Components

SUMMARY:
The primary purpose of this study is to demonstrate cumulative revision rate of the REDAPT System Monolithic Sleeveless/Sleeved Stem, Fully Porous Acetabular Shell with XLPE liner, and Modular Shell Components (with or without Staple, Slice and Blade Augments) at 10 years.

DETAILED DESCRIPTION:
Retrospective-prospective, single arm, multicenter study of subjects previously implanted with the REDAPT System Monolithic Sleeveless/Sleeved Stem and/or Fully Porous Acetabular Shell with XLPE liner and/or Modular Shell Components (with or without Staple, Slice and Blade Augments).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to enroll in the study:

1. Subject was considered skeletally mature at the time of surgery and was at least 18 years of age.
2. Subject has undergone hip arthroplasty with the REDAPT Fully Porous Acetabular Shell with XLPE liner or REDAPT Modular Cup Components (with or without Staple, Slice and Blade Augments), and/or Monolithic Sleeveless Stem, and/or Monolithic Sleeved Stem and are at least 3 months post-implantation at this site.
3. Subject required surgery with REDAPT device chosen for one of the following indications:

   1. Advanced degeneration of the hip joint as result of osteoarthritis, avascular necrosis, posttraumatic arthritis, rheumatoid arthritis, or dysplasia (or any of the composites of these conditions).
   2. Fracture-dislocation of the hip, femoral neck fracture or trochanteric fractures of the proximal femur with head involvement that are unmanageable using other techniques.
   3. Revision THA
4. Subject is willing to consent to and to follow the study visit schedule (as defined in the study protocol and ICF), by signing the IRB/IEC approved ICF.
5. Subject is willing and able to participate in required follow-up visits at the investigational site and to complete study procedures.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be excluded from study participation:

1. Subject had an active infection - systemic or at the site of surgery.
2. Subject, in the opinion of the PI, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
3. Subject is known to be at risk for loss to follow-up or failure to return for scheduled visits.
4. Subject is incarcerated or is pending incarceration.
5. Subject is enrolled in another clinical study that would affect the endpoints of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject has undergone hip arthroplasty with the REDAPT Fully Porous Acetabular Shell with XLPE liner or REDAPT Modular Cup Components (with or without Staple, Slice and Blade Augments), and/or Monolithic Sleeveless Stem, and/or Monolithic Sleeved Stem and are at least 3 months post-implantation at this site.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2034-07-01 (Estimated); Study Completion 2034-07-01 (Estimated)

PRIMARY OUTCOMES:
Revision rate | 10 years post-op
  REDAPT System Monolithic Sleeveless/Sleeved Stem, Fully Porous Acetabular Shell with XLPE liner and Modular Shell Components (with or without Staple, Slice and Blade Augments) cumulative revision rate for any reason 10 years postoperatively.

SECONDARY OUTCOMES:
EuroQul Five Dimensions Questionnaire EQ-5D-5L | Collect retrospectively from medical records preoperatively and at 1 year, and prospectively at 2, 5, and 10 years post-operatively
  Clinical evaluation to assess changes over time from pre-op through 10 years post-op. The EuroQol Five Dimensions (EQ-5D) Questionnaire is an instrument that derives a single index for Quality of Life (QoL) and has two sections. The first section consists of five questions covering the dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The second part consists of a 20-centimeter vertical VAS ranging from 0 to 100. It records the respondent's self-rated health where the endpoints are labeled 'Best imaginable health state' and 'Worst imaginable health state'. EQ-5D-5L is completed by the subject.
Functional outcomes as determined by the Hip Disability Osteoarthritis Outcome (HOOS) score | Collect retrospectively from medical records preoperatively and at 1 year, and prospectively at 2, 5, and 10 years post-operatively
  HOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related QOL. The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Radiographic assessments | Collect retrospectively from medical records preoperatively and at 1 year, and prospectively at 2, 5, and 10 years post-operatively
  Loosening as indicated by radiolucencies (RLL) > 2mm; Lack of evidence of surface wear or particulate debris generation as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Nahomie Prophete, Study Chair — Smith & Nephew, Inc.
Locations (4):
- United States (4):
  - Eisenhower Medical Center-Hospital, Rancho Mirage, California
  - Scripps Mercy, San Diego, California
  - NYU Langone Health Orthopedic Hospital, New York, New York
  - Hospital for Surgery- New York, New York, New York